CLINICAL TRIAL: NCT02546258
Title: A Prospective, Open Label, Non-comparative Clinical Investigation to Evaluate the Performance of a Fungal Nail Treatment on the Visual Signs of Onychomycosis
Brief Title: Evaluation of the Performance of a Fungal Nail Treatment on the Visual Signs of Onychomycosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Reckitt Benckiser Healthcare (UK) Limited (Industry)
Collaborators: Intertek (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NPD810
Record Dates: First submitted 2015-09-08; First posted 2015-09-10 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2015-11

CONDITIONS: Onychomycosis of Toenails
Keywords: Fungal Nail

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A Funagl Nail Treatment (Other): Marketed treatment of Fungal Nail Follow instructions on pack
  Interventions: Device: A Fungal Nail Treatment

INTERVENTIONS:
Device: A Fungal Nail Treatment — treats the signs of mild fungal nail infections
  Other Names: Funagl Nail Treatment

SUMMARY:
This is a prospective, open label, non-comparative clinical investigation to evaluate the performance of a Fungal Nail Treatment on the visual signs of onychomycosis.

The Fungal Nail Treatment is a CE Marked Class I Medical Device and is commercially available as an over-the-counter product.

The ability of the Fungal Nail Treatment to treat the visual signs of mild fungal toenail infections will be determined by a reduction in the surface area of the infection over time. This will be assessed through visual quantification of the infected area from baseline, as measured by image analysis, throughout the treatment period, where subjects will follow instructions for use on the product pack and self-treat for the duration of the investigation or until their condition has resolved. Both subject and podiatrist will assess the improvement of signs and symptoms of the target nail.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent has been obtained.
* Age between 18 years to 65 years inclusive.
* Gender: male and female subjects.
* Subjects with visual signs of MILD fungal nail infection present on at least one big toenail or with fungal nail infection on one other toenail on the same foot, in addition to the target big toenail (condition of other foot not relevant) as per podiatrist visual assessment.
* Subjects with no more than 50% surface area of the target big toenail visually affected, from the leading distal edge, as assessed by the podiatrist.

Exclusion Criteria:

* Subjects with moderate to severe fungal toenail infection, on either big toenail, as determined by podiatrist assessment.
* Subjects with fungal nail infection on more than two toenails on their target foot.
* Subjects reporting presence of visual symptoms of fungal toenail infection for more than five years.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-08-25 (Actual); Primary Completion 2014-11-21 (Actual); Study Completion 2014-11-21 (Actual)

PRIMARY OUTCOMES:
Percentage reduction of the surface area of infection over time using image analysis | 40 weeks

SECONDARY OUTCOMES:
Percentage reduction of the surface area of infection over time from baseline to week 4 using image analysis | 4 weeks
The proportion of subjects whose fungal nail infection has resolved | 40 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rashid Haye, MBBS MD, Principal Investigator — Intertek CRS
Locations (1):
- Intertek CRS, Manchester, United Kingdom